CLINICAL TRIAL: NCT05234320
Title: A Phase 1, Randomized, Double-blinded, Vehicle-controlled, Single and Multi-Dose, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Volunteers of the Novel Self-Administered Intranasal CG- SpikeDown Antiviral Drug
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Volunteers of the Novel Self-Administered Intranasal CG- SpikeDown Antiviral Drug
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Caregen Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CG-S-P01
Record Dates: First submitted 2022-02-06; First posted 2022-02-10 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A Phase 1, Randomized, Double-blinded, Vehicle-controlled, Single and Multi-Dose, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics
Who Masked: Outcomes Assessor
Masking Description: The study will begin with recruitment for the single 25 mg dose arm /vehicle arm, and once all subjects have been treated and attended their first follow-up visit with no significant safety issues, recruitment of participants for the single 50 mg dose arm/vehicle arm and the multiple 25 mg dose arm/vehicle arm. Once subjects from the multi 25 mg dose Cohort have attended their follow-up visit with no significant safety issues, recruitment for the final multiple 50 mg dose arm/vehicle arm may commence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- stage I- Healty (Experimental): The first 2 patients in this stage will receive the vehicle treatment and will not undergo the first 24 hour hospitalization. The 3rd and 4th patients will receive a lower dose of 12.5 mg of the DP once daily for 7 days, and the first 24 hours will be hospitalized for the first 24 hours. The 5th patient will receive the 25 mg from the DP once daily for 7 days and will be hospitalized for the first 24 hours. The next 2 patients will receive the 25 mg dose and will not undergo the first 24 hour hospitalization. The next 3 patients will receive the optimal dose of 50 mg and will not undergo the first 24 hour hospitalization
  Interventions: Drug: CG-SpikeDown, intranasal formulation
- Stage II- Placebo + SOC (Active Comparator): This arm will be include 20 This arm will be include 20 symptomatic non-hospitalized COVID-19 patients and will be conducted at patients' homes during their self-isolation, and they will be received Placebo + standard of care
  Interventions: Drug: Vehicle (Placebo); Drug: Standard of core (type of therapy is depend of decide of the site)
- Stage II- DP low dose (25 mg) + SOC (Active Comparator): This arm will be include 20 symptomatic non-hospitalized COVID-19 patients and will be conducted at patients' homes during their self-isolation, and they will be received Drug product low does(25 mg) + standard of care
  Interventions: Drug: CG-SpikeDown, intranasal formulation; Drug: Vehicle (Placebo); Drug: Standard of core (type of therapy is depend of decide of the site)
- Stage II- DP planned dose (50 mg) + SOC (Active Comparator): This arm will be include 20 This arm will be include 20 symptomatic non-hospitalized COVID-19 patients and will be conducted at patients' homes during their self-isolation, and they will be received Drug product planned does(50 mg) + standard of care
  Interventions: Drug: CG-SpikeDown, intranasal formulation; Drug: Vehicle (Placebo); Drug: Standard of core (type of therapy is depend of decide of the site)

INTERVENTIONS:
Drug: CG-SpikeDown, intranasal formulation — The CG-SpikeDown peptide produces a dose-dependent increase in binding to the receptor binding domain (RBD) of the SARS-CoV-2 spike protein and a dose-dependent inhibition of SARS-CoV-2 protein binding to ACE2, the key cellular target. A similar inhibition of binding to ACE2 in human alveolar basal epithelial cells has been demonstrated.
  Arms: Stage II- DP low dose (25 mg) + SOC; Stage II- DP planned dose (50 mg) + SOC; stage I- Healty
Drug: Vehicle (Placebo) — patients will receive active drug or placebo in addition to standard of care
  Arms: Stage II- DP low dose (25 mg) + SOC; Stage II- DP planned dose (50 mg) + SOC; Stage II- Placebo + SOC
Drug: Standard of core (type of therapy is depend of decide of the site) — patients will receive active drug or placebo in addition to standard of care
  Arms: Stage II- DP low dose (25 mg) + SOC; Stage II- DP planned dose (50 mg) + SOC; Stage II- Placebo + SOC

SUMMARY:
Study Design This is a phase 1, randomized, Vehicle-controlled, double-blinded study to assess the safety of Caregen Intranasal CG-SpikeDown in healthy subjects.

All randomized subjects will receive an active drug or Vehicle. Subjects randomized to the DP(Drug product) active treatment will receive CG- SpikeDown intranasally once daily for one or seven days at either a low (25 mg) or planned (50 mg) dose.

Subject recruitment will be conducted via study advertisement on social media, and subjects will be adequately compensated. The subjects will arrive each day at the clinic to receive the treatment and will be hospitalized for safety monitoring for the first 24 hours post-DP or vehicle administration.

DETAILED DESCRIPTION:
This is a phase 1, Randomized, Double-blinded, Vehicle-controlled, Single and Multi-Dose, Dose Escalation Study, which will assess the safety of the Caregen CG-SpikeDown drug self-administered intranasally, for healthy subjects.

The study will include 16 healthy subjects and will be conducted in a clinic under complete supervision of the clinical team. The study will start with evaluation of the lowest dose, that will be increased gradually as long as no safety issues arise.

At the first stage of the study, three (3) subjects will be randomized in a 1:2 ratio to receive vehicle treatment or the active drug, respectively. Each of the 3 subjects will receive a single 25 mg dose of the assigned treatment. These subjects will be referred as Cohort 1. If no safety issues arise, the study will proceed simultaneously to the second and third stages, as depicted in Figure 1 Study Flow Chart.

At the second stage of the study, additional three (3) subjects will be enrolled and randomized in a 1:2 ratio to receive vehicle treatment or the active drug, respectively. Each of the 3 subjects will receive a single 50 mg dose of the assigned treatment. These subjects will be referred as Cohort 2. If no safety issues arise, the study will proceed to the 4th stage.

At the third stage of the study, additional three (5) subjects will be enrolled. The first 2 subjects (out of the 5 subjects) will receive an open label DP treatment-a daily 25 mg dose for 7 days. The open-label subjects will undergo PK assessments as described in the SOA. The next 3 subjects will be randomized in a 1:2 ratio to receive vehicle treatment or the active drug, respectively. Each of the 3 subjects will receive a daily 25 mg dose of the assigned treatment for 7 days. These subjects will be referred as Cohort 3.

At the fourth stage of the study, additional three (5) subjects will be enrolled. The first 2 subjects (out of the 5 subjects) will receive an open label DP treatment-a daily 50 mg dose for 7 days. The open-label subjects will undergo PK assessments as described in the SOA. The next 3 subjects will be randomized in a 1:2 ratio to receive vehicle treatment or the active drug, respectively. Each of the 3 subjects will receive a daily 50 mg dose of the assigned treatment for 7 days. These subjects will be referred as Cohort 4.

The main objective of this study is to assess the toxicity and the pharmacokinetic (PK) parameters of the Drug Product (DP). Subjects will be recruited to the study via study advertisement on social media and the subjects will be adequately compensated. The DP will be self-administered intranasally once daily for 1 day or seven days, depending on the study cohort. PK parameters will be evaluated for 4 subjects participating in the 7 daily DP doses study cohorts. Blood samples for this purpose will be collected at several time points (as described in SOA) during Day 1 and Day 7 of treatment. Toxicity will be evaluated during the entire study period.

Patients receiving a single dose will arrive for a follow-up visit 72 hours following DP administration (24 hours following hospital discharge), again 7 days (+-2 days) following DP administration, and again 14 days (+-2 days) following DP administration. Subjects receiving a daily dose for 7 days will be followed up 14 days (+-2 days) following initial DP administration (7 days (+-2 days) following final DP administration).

Safety review by the DSMB will occur following treatment of the last subject in each study arm.

ELIGIBILITY:
Stage I Inclusion Criteria

1. Age ≥ 18 years in healthy condition
2. Able and willing to sign ICF

Stage I Exclusion Criteria

1. Known hypersensitivity to any of the DP ingredients.
2. Pregnant or lactating woman.
3. Participation in another clinical study within 4 weeks from screening
4. Patient has a positive test for HBV, HCV or HIV
5. Subjects diagnosed with allergic rhinitis and/or deviated septum and/or sinusitis.
6. Any medical condition that in the investigator's opinion will jeopardize the patient's ability to follow the protocol.

Stage II Inclusion Criteria

1. Age ≥ 18 years
2. Laboratory confirmed SARS-CoV2 Infection by nasopharyngeal RT-PCR.
3. COVID-19 symptoms within 3 days of symptoms onset
4. Patients diagnosed with COVID-19 that are not hospitalized (classified on the NIAID 8-point ordinal scale as 1 or 2).

Stage II Exclusion Criteria

1. Patients who may require hospitalization during the study
2. Immunocompromised COVID-19 patients.
3. Known hypersensitivity to any of the DP ingredients.
4. Patient has a positive test for HBV, HCV or HIV
5. Pregnant or lactating woman.
6. Participation in another clinical study within 4 weeks from screening
7. Subjects diagnosed with allergic rhinitis and/or deviated septum and/or sinusitis.
8. Any medical condition that in the investigator's opinion will jeopardize the patient's ability to follow the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
SARS Cov-2 RT-PCR test | 7 days
  Viral load is estimated from nasopharyngeal swabs and instructions for use is based on the package insert of the diagnostic. This assessment will be used to diagnose COVID-19 patients during Stage II in case they do not have a positive COVID-19 test result from 72 hours before the Stage II screening visit, and will also be used to assess viral load in COVID-19 patients during Stage II.
Area under the plasma concentration versus time curve | 7 days
  The following PK parameters evaluation collected 10 minutes prior to DP self-administration, immediately following DP self-administration, and 1, 2, 4 and 6 hours following DP self-administration, on Day 1 and Day 6 of treatment. These measurements will be collected only during Stage I (from 10 healthy subjects)

SECONDARY OUTCOMES:
NIAID ordinal scale | 14 days
  Time to sustained clinical recovery. Sustained clinical recovery will be defined based on self-reported key COVID-19 related symptoms using the NIAID ordinal scale.
  • Clinical status on Day 7 and Day 14 assessed on the NIAID 8-point ordinal scale consisting of the following categories:
  1. Not hospitalized, no limitations on activities;
  2. Not hospitalized, limitation on activities and/or requiring home oxygen;
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  5. Hospitalized, requiring supplemental oxygen;
  6. Hospitalized, on noninvasive ventilation or high-flow oxygen devices;
  7. Hospitalized, on invasive mechanical ventilation or ECMO; and
  8. Death
  Maximum is 1. Not hospitalized, no limitations on activities; Minimum is 8. Death
Peak Plasma Concentration | 7 days
  The following PK parameters evaluation collected 10 minutes prior to DP self-administration, immediately following DP self-administration, and 1, 2, 4 and 6 hours following DP self-administration, on Day 1 and Day 6 of treatment. These measurements will be collected only during Stage I (from 10 healthy subjects)

OTHER OUTCOMES:
Time to maximum plasma concentration | 7 days
  The following PK parameters evaluation collected 10 minutes prior to DP self-administration, immediately following DP self-administration, and 1, 2, 4 and 6 hours following DP self-administration, on Day 1 and Day 6 of treatment. These measurements will be collected only during Stage I (from 10 healthy subjects)

IPD SHARING:
Plan to Share IPD: No